CLINICAL TRIAL: NCT05742503
Title: Effects of Different Progesterone Containing Contraceptive Methods on Safety and Endogenous Progesterone Level
Brief Title: Progesterone Containing Contraceptive Methods on Endogenous Progesterone Level
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Ossman, Assistant Professor of Obstetrics and Gynecology Department,Faculty of Medicine,Tanta University, Tanta University
Other Study IDs: 36035/11/22
Record Dates: First submitted 2022-12-15; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Progesterone; Contraceptive Methods
MeSH Terms: interventions — Medroxyprogesterone Acetate; etonogestrel; Norgestrel; Levonorgestrel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Depo-Provera group: This group will receive150 mg of injectable progesterone every 90 days or 3 months
  Interventions: Other: Depo-Provera
- Implanon group: This group will receive 68 mg of etonogestrel implant formerly known as Implanon.
  Interventions: Other: Implanon
- Norgestrel group: This group will receive 0.075 mg of norgestrel (Ovrette®) once daily.
  Interventions: Other: Norgestrel
- Mirena group: This group will receive IUD (Mirena) containing 52 mg of levonorgestrel.
  Interventions: Other: Mirena

INTERVENTIONS:
Other: Depo-Provera — Injectable progesterone
  Groups: Depo-Provera group
Other: Implanon — Etonogestrel implant
  Groups: Implanon group
Other: Norgestrel — Pill containing progesterone
  Groups: Norgestrel group
Other: Mirena — Levonorgestrel-releasing intra-uterine drug (IUD)
  Groups: Mirena group

SUMMARY:
The aim of this study is to assess the effect of different progesterone containing contraceptive methods on safety and endogenous progesterone level

DETAILED DESCRIPTION:
Progestogen-only' contraceptives are presented as injections, implants, oral formulations, hormone-releasing intrauterine methods and emergency contraceptives. These substances could be used by females who are breastfeeding or have other contraindications to estrogen treatment, including those who are immediately postpartum, have thalassemia, sickle-cell disease, gallbladder disease, or currently experiencing thrombo-embolic disorders, valvular heart disease, ischemic heart disease.

Intrauterine, injectable methods and contraceptive implants named as long-acting reversible contraceptives (LARC) are the more efficient reversible contraceptive approaches are highly effective, longer-acting contraceptive methods levels.

ELIGIBILITY:
Inclusion Criteria:

* 80 healthy fertile females
* 20-35 years
* With normal menstrual history
* Had at least one offspring after spontaneous pregnancy

Exclusion Criteria:

* Any disease affects uterus (uterine tumors fibroids, endometriosis, prolapse, or tuberculosis).
* Ovarian tumors
* submucous myoma
* irregular menstrual cycle
* past or family history of breast disease
* Diabetic patients,
* medication affecting reproductive or metabolic functions.
* endometrial thickness <7 mm on the secretory transformation day
* history of spontaneous abortions
* history of embryo transfer failure on over three occasions
* Patients had cortisol medications
* patients who received radiological treatment

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Among patients attending Tanta University Hospitals
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Assess the effect of different progesterone containing contraceptive methods on safety and endogenous progesterone level | Six mounths
  The effect of different progesterone containing contraceptive methods on safety and endogenous progesterone level will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Mona K Omar, MD, Principal Investigator — Assistant Professor of Obstetrics and Gynecology Department, Faculty of Medicine,Tanta University
Locations (1):
- Ahmed Ossman, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the principal investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: One year